CLINICAL TRIAL: NCT02144766
Title: Prevention of Pro-inflammatory Cytokines-associated Myocardial Dysfunction and Injury Resulting From Salter Innominate Osteotomy by Caudal Block
Brief Title: Prevention of Myocardial Dysfunction and Injury Resulting From Salter Innominate Osteotomy by Caudal Block
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Si-Qin Chen (Other)
Responsible Party: Sponsor-Investigator, Si-Qin Chen, attending doctor, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 060717
Record Dates: First submitted 2014-05-11; First posted 2014-05-22 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Cardiac Dysfunction; Myocardial Injury
MeSH Terms: interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ropivacaine (Experimental): caudal block with 1 ml/kg of ropivacaine 0.2%
  Interventions: Drug: ropivacaine
- saline (Placebo Comparator): caudal block with 1 ml/kg of saline
  Interventions: Drug: saline

INTERVENTIONS:
Drug: ropivacaine — caudal block with 1 ml/kg of ropivacaine 0.2%
  Arms: Ropivacaine
Drug: saline — caudal block with 1 ml/kg of saline
  Arms: saline

SUMMARY:
The goal of the present study was to investigate the role of pro-inflammatory cytokines in myocardial dysfunction and injury resulting from noncardiac injury in children and whether or not anti-inflammatory treatment with caudal block prevents pro-inflammatory cytokines-associated myocardial dysfunction and injury following noncardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed for developmental dysplasia of the hip (DDH) undergoing Salter innominate osteotomy will be recruited into the study.

Exclusion Criteria:

* Children with anemia, electrolyte disturbances, abnormal acid-base status, bleeding diathesis, history of allergy to local anesthetics, neurologic and spinal diseases, skin infections on the caudal area, renal dysfunction, symptomatic cardiovascular and respiratory disease

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2014-04; Primary Completion 2014-09 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
change from baseline(before induction of anesthesia) in plasma concentrations of NT(N terminal)-proBNP at arrival in the postanesthesia care unit | baseline(before induction of anesthesia), arrival in the postanesthesia care unit
change from baseline(before induction of anesthesia) in plasma concentrations of NT(N terminal)-proBNP at 3h after surgery | baseline(before induction of anesthesia), 3h after surgery
change from baseline(before induction of anesthesia) in plasma concentrations of NT(N terminal)-proBNP at 24h after surgery | baseline(before induction of anesthesia), 24h after surgery
change from baseline(before induction of anesthesia) in plasma concentrations of NT(N terminal)-proBNP at 48h after surgery | baseline(before induction of anesthesia), 48h after surgery
change from baseline(before induction of anesthesia) in plasma concentrations of NT(N terminal)-proBNP at 72h after surgery | baseline(before induction of anesthesia), 72h after surgery
change from baseline(before induction of anesthesia) in plasma concentrations of CK(creatine kinase)-MB at arrival in the postanesthesia care unit | baseline(before induction of anesthesia), arrival in the postanesthesia care unit
change from baseline(before induction of anesthesia) in plasma concentrations of CK(creatine kinase)-MB at 3h after surgery | baseline(before induction of anesthesia), 3h after surgery
change from baseline(before induction of anesthesia) in plasma concentrations of CK(creatine kinase)-MB at 24h after surgery | baseline(before induction of anesthesia), 24h after surgery
change from baseline(before induction of anesthesia) in plasma concentrations of CK(creatine kinase)-MB at 48h after surgery | baseline(before induction of anesthesia), 48h after surgery
change from baseline(before induction of anesthesia) in plasma concentrations of CK(creatine kinase)-MB at 72h after surgery | baseline(before induction of anesthesia), 72h after surgery
change from baseline(before induction of anesthesia) in plasma concentrations of cTn(troponin)I at arrival in the postanesthesia care unit | baseline(before induction of anesthesia), arrival in the postanesthesia care unit
change from baseline(before induction of anesthesia) in plasma concentrations of cTn(troponin)I at 3h after surgery | baseline(before induction of anesthesia), 3h after surgery
change from baseline(before induction of anesthesia) in plasma concentrations of cTn(troponin)I at 24h after surgery | baseline(before induction of anesthesia), 24h after surgery
change from baseline(before induction of anesthesia) in plasma concentrations of cTn(troponin)I at 48h after surgery | baseline(before induction of anesthesia), 48h after surgery
change from baseline(before induction of anesthesia) in plasma concentrations of cTn(troponin)I at 72h after surgery | baseline(before induction of anesthesia), 72h after surgery
change from baseline(before induction of anesthesia) in plasma concentrations of TNF(tumor necrosis factor)-α at arrival in the postanesthesia care unit | baseline(before induction of anesthesia), arrival in the postanesthesia care unit
change from baseline(before induction of anesthesia) in plasma concentrations of TNF(tumor necrosis factor)-α at 3h after surgery | baseline(before induction of anesthesia), 3h after surgery
change from baseline(before induction of anesthesia) in plasma concentrations of TNF(tumor necrosis factor)-α at 24h after surgery | baseline(before induction of anesthesia), 24h after surgery
change from baseline(before induction of anesthesia) in plasma concentrations of TNF(tumor necrosis factor)-α at 48h after surgery | baseline(before induction of anesthesia), 48h after surgery
change from baseline(before induction of anesthesia) in plasma concentrations of TNF(tumor necrosis factor)-α at 72h after surgery | baseline(before induction of anesthesia), 72h after surgery
change from baseline(before induction of anesthesia) in plasma concentrations of IL(interleukin)-6 at arrival in the postanesthesia care unit | baseline(before induction of anesthesia), arrival in the postanesthesia care unit
change from baseline(before induction of anesthesia) in plasma concentrations of IL(interleukin)-6 at 3h after surgery | baseline(before induction of anesthesia), 3h after surgery
change from baseline(before induction of anesthesia) in plasma concentrations of IL(interleukin)-6 at 24h after surgery | baseline(before induction of anesthesia), 24h after surgery
change from baseline(before induction of anesthesia) in plasma concentrations of IL(interleukin)-6 at 48h after surgery | baseline(before induction of anesthesia), 48h after surgery
change from baseline(before induction of anesthesia) in plasma concentrations of IL(interleukin)-6 at 72h after surgery | baseline(before induction of anesthesia), 72h after surgery

SECONDARY OUTCOMES:
change from baseline(just before the start of surgery) in MAP(mean arterial pressure) at arrival in the postanesthesia care unit | baseline(just before the start of surgery), at arrival in the postanesthesia care unit
change from baseline(just before the start of surgery) in MAP(mean arterial pressure) at 3h after surgery | baseline(just before the start of surgery), 3h after surgery
change from baseline(just before the start of surgery) in CVP(central venous pressure) at arrival in the postanesthesia care unit | baseline(just before the start of surgery), at arrival in the postanesthesia care unit
change from baseline(just before the start of surgery) in CVP(central venous pressure) at 3h after surgery | baseline(just before the start of surgery), 3h after surgery
change from baseline(just before the start of surgery) in HR(heart rate) at arrival in the postanesthesia care unit | baseline(just before the start of surgery), at arrival in the postanesthesia care unit
change from baseline(just before the start of surgery) in HR(heart rate) at 3h after surgery | baseline(just before the start of surgery), 3h after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhua Hospital, Shanghai, China